CLINICAL TRIAL: NCT03849781
Title: Enhanced Heart Rate Monitoring of Newborns After Birth and During Resuscitation
Brief Title: The NeoBeat Efficacy Study for Newborns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Sykehuset Østfold (Unknown); Laerdal Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SUS2019SIR
Record Dates: First submitted 2019-01-30; First posted 2019-02-21 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-01

CONDITIONS: Newborn Resuscitation; Heart Rate Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): NeoBeat will be placed on all newborns immediately after birth to assess the heartrate for at least 5 minutes, or longer if the newborn needs resuscitation. Intervention subjects will have a visible display of the heart rate on the NeoBeat, to guide healthcare providers in further management of the newborn.
  Interventions: Device: NeoBeat with a visible display
- Standard Care (No Intervention): NeoBeat will be placed on the newborn to collect information on heart rate, but heart rate is not displayed to the healthcare providers. If the newborn is in need of resuscitation to initiate spontaneous respiration, the baby will be transferred to the resuscitation bay. According to recommendations the heart rate should be assessed and positive pressure ventilation initiated within one minute of life. Standard care is to assess heart rate by conventional ECG and/or pulse oximetry, alternatively auscultation of the heart.

INTERVENTIONS:
Device: NeoBeat with a visible display — NeoBeat (Laerdal Medical) is a CE approved novel heart rate meter, able to detect heart rate in newborns within seconds of birth. The NeoBeat uses ECG dry-electrodes in a snug-fit abdomen-shaped buckle for rapid application around the newborn's abdomen or thorax. It allows healthcare providers to reliably assess heart rate of the newborn immediately after birth and continuously during resuscitation.
  Arms: Intervention

SUMMARY:
In a multicenter randomized controlled trial the investigators will evaluate the efficacy of the novel heart rate meter NeoBeat on ventilation performance and short-term outcomes compared to standard care in newborns in need of positive pressure ventilation to initiate spontaneous breathing after birth.

DETAILED DESCRIPTION:
Heart rate assessment immediately after birth in newborn infants is the most important clinical indicator to evaluate the status of a newborn, and critical to the correct guidance of resuscitation efforts.

One of the knowledge gaps identified by the International Liason Committee on Resuscitation (ILCOR) is how best to assess ventilation during newborn resuscitation, and improved technology for rapid application of ECG.

Laerdal Medical has developed a novel heart rate meter, NeoBeat, implementing ECG dry-electrodes in a snug-fit abdomen-shaped buckle for for rapid application on the newborn.

In a multicenter randomized controlled trial the investigators will study the efficacy of NeoBeat on ventilation performance and short-term outcomes compared to standard care in newborns in need of positive pressure ventilation to initiate spontaneous respiration after birth.

ELIGIBILITY:
Inclusion Criteria:

Inborn, Gestational age ≥ 28 weeks, Multiples according to availability of equipment

Exclusion Criteria:

Congenital malformations that interfere with the intervention, Non-consent

Max Age: 60 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2019-03-08 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of cases with adherence to resuscitation guidelines in non-breathing newborns | First minute after birth
  Defined as initiation of PPV within on minute

SECONDARY OUTCOMES:
Change in time from birth to initiation of PPV | first 15 minutes of life
  defined as seconds between birth and initiation of PPV
Change in total duration of PPV | first hour of life
  defined as seconds of PPV in total
Change in time from birth to a stable HR ≥100 and 120 bpm | first hour of life
  defined as HR ≥100 and 120 bpm for ≥ 60 seconds after discontinuing PPV
Change in time for pulse oximeter saturation to reach stable values of ≥ 95% without oxygen supplementation | first hour of life
  defined as seconds between birth to reach saturation values ≥ 95% without oxygen supplementation
Adequate Vt delivered during PPV | first hour of life
  defined as proportion of time of PPV with Vt ≥ 6 ml/kg
Change in ventilation fraction | first hour of life
  defined as cumulative number of seconds with PPV efforts excluding pauses
Change in number of infants with Apgar score <7 at 5 and 10 minutes | first 10 minutes of life
  Apgar score at 5 and 10 minutes
Change in NICU admission rate after resuscitation | first hour of life
  defined as percentage of newborns needing admission to the NICU after resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Svein Skeie, MD PhD, Study Director — Stavanger University Hosptial
Locations (1):
- Stavanger University Hospital, Stavanger, Rogaland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rettedal S, Kibsgaard A, Kvaloy JT, Eilevstjonn J, Ersdal HL. Prevalence of bradycardia in 4876 newborns in the first minute after birth and association with positive pressure ventilation: a population-based cross-sectional study. Arch Dis Child Fetal Neonatal Ed. 2024 Jun 19;109(4):371-377. doi: 10.1136/archdischild-2023-325878. PMID 37940377
- [Derived] Rettedal S, Kibsgaard A, Eilevstjonn J, Kvaloy JT, Bjorland PA, Markhus Pike H, Haynes J, Tysland TB, Stordal K, Holte K, Davis PG, Ersdal HL. Impact of immediate and continuous heart rate feedback by dry electrode ECG on time to initiation of ventilation after birth: protocol for a randomised controlled trial. BMJ Open. 2022 Sep 7;12(9):e061839. doi: 10.1136/bmjopen-2022-061839. PMID 36691167